CLINICAL TRIAL: NCT02048657
Title: The Efficiency of ProSeal Laryngeal Mask Airway Insertion: Compared the Techniques of Foley Airway Stylet Tool With Introducer-Tool
Brief Title: The Effectiveness of Foley Airway Stylet Tool on Proseal LMA Insertion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KMHK-IRB-96023
Record Dates: First submitted 2013-10-23; First posted 2014-01-29 (Estimated); Last update posted 2014-01-29 (Estimated); Status verified 2008-03

CONDITIONS: Anesthesia Insertion Complication; Airway Morbidity
Keywords: LMA, Foley Airway Stylet Tool (FAST), introducer-tool (I-Tool)
MeSH Terms: conditions — Fasting

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Foley group (Experimental): The Foley Airway Stylet Tool was used to guide ProSeal LMA insertion
  Interventions: Device: Foley Airway Stylet Tool
- I-Tool group (Experimental): the ProSeal LMA was inserted with a standard introducer-tool
  Interventions: Device: introducer-tool

INTERVENTIONS:
Device: Foley Airway Stylet Tool
  Arms: Foley group
Device: introducer-tool
  Arms: I-Tool group

SUMMARY:
Due to its soft cuff easily folded to impede ProSeal LMA insertion, many tools are developed. The aim of the study is to investigate the efficiency of ProSeal LMA insertion guided by a soft, direct optical Foley airway stylet tool (FAST) and compared with the standard introducer-tool (I-Tool).

ELIGIBILITY:
Inclusion Criteria:

1. patients with American Society of Anesthesiologists physical status I-II
2. aged 20-65 years
3. requiring LMA Intubation under general anesthesia
4. unlimited mouth open
5. unlimited neck motion

Exclusion Criteria:

1. mouth open < 3 cm
2. limited neck motion
3. BMI≧35 kg/m2

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2008-03; Primary Completion 2009-03 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Number of participants with successful airway establishment | half an hour
  successful airway establishment is defined as adequate ventilation with ProSeal LMA and its alignment with viewing of proper glottic and esophageal positions.

SECONDARY OUTCOMES:
postoperative sore throat | 2 days
  sore throat recorded in recovery room and in the coming morning
hoarseness | 2 days
  severity of hoarseness was recorded in recovery room and in the coming morning

CONTACTS AND LOCATIONS:
Overall Officials: Kuang I Cheng, MD, PhD., Study Director — Department of anesthesiology, Kaohsiung Medical University, Taiwan
Locations (1):
- Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City, Kaohsiung, Taiwan

REFERENCES:
- [Derived] Chen MK, Hsu HT, Lu IC, Shih CK, Shen YC, Tseng KY, Cheng KI. Techniques for the insertion of the ProSeal laryngeal mask airway: comparison of the Foley airway stylet tool with the introducer tool in a prospective, randomized study. BMC Anesthesiol. 2014 Nov 18;14:105. doi: 10.1186/1471-2253-14-105. eCollection 2014. PMID 25435806